CLINICAL TRIAL: NCT06056804
Title: Efficacy and Safety of Neoadjuvant Chemoradiotherapy Combined With PD-1 Inhibitor and Thymalfasin in pMMR/MSS Locally Advanced Middle and Low Rectal Cancer: An Open, Multi-center, Prospective, Single-arm Phase II Clinical Study
Brief Title: Neoadjuvant Chemoradiotherapy Combined With PD-1 Inhibitor and Thymalfasin for pMMR/MSS Locally Advanced Mid-low Rectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZDX+PD-1-LARC
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-08

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: pMMR/MSS; locally Advanced Rectal Cancer; PD-1; neoadjuvant; chemoradiation; Thymalfasin
MeSH Terms: interventions — Capecitabine; tislelizumab; Thymalfasin

STUDY DESIGN:
Intervention Model Description: neoadjuvant chemoradiotherapy combined with PD-1 monoclonal antibody and thymalfasin
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cCRT+tislelizumab+thymalfasin (Experimental): A total of 20 pMMR/MSS locally advanced middle and low rectal cancer patients will receive long-course concurrent chemoradiotherapy combined with 3 cycles of tislelizumab and 11 weeks of thymalfasin therapy.
  Interventions: Drug: capecitabine; Drug: tislelizumab; Drug: thymalfasin; Radiation: long-term radiotherapy

INTERVENTIONS:
Drug: capecitabine — 825-1000mg/m2,po,bid
Drug: tislelizumab — 200mg,iv.gtt,q3w
Drug: thymalfasin — 4.8mg,sc,biw
Radiation: long-term radiotherapy — 50 Gy/25 f, 2 Gy/day

SUMMARY:
This is an open, prospective, multi-center, single-arm phase II clinical study assessing the efficacy and safety of neoadjuvant chemoradiotherapy combined with PD-1 inhibitor and thymalfasin in patients with pMMR/MSS locally advanced middle and low rectal cancer.

DETAILED DESCRIPTION:
This study is an open, prospective, multi-center, single-arm phase II clinical study. In this study, patients with pMMR/MSS locally advanced middle and low rectal cancer were selected as the subjects and treated with neoadjuvant treatment protocol of long-course concurrent chemoradiotherapy combined with PD-1 monoclonal antibody and thymalfasin. The primary endpoint of the study was complete response (CR) rate. The secondary end points included treatment-related adverse events (TRAEs) rate, 30-day incidence of postoperative complications, objective response rate (ORR), 3-year disease-free survival (DFS) rate, Neoadjuvant rectal cancer (NAR) score, R0 resection rate, and anal preservation rate.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were fully informed of the study and voluntarily signed the informed consent form;
2. Patients with rectal cancers must satisfied all the following conditions:

1) Stage II/III LARC (cT3-4aN0M0 and cT1-4aN1-2M0); 2) Tumor distal located ≤ 10 cm from anal verge (MRI diagnosed); 3) pMMR or MSS confirmed by immunohistochemistry or genetic test. 3.Patients regardless of gender with aged ≥18 years and ECOG score of 0 or 1; 4. Physical and viscera function of patients can withstand major abdominal surgery; 5.Patients are willing and able to follow the study protocol during the study 6.Patients give consent to the use of pathological specimens for study 7.Within 28 days prior to enrolment, we must confirm a negative serological pregnancy test for child-bearing age women and they agree to use effective contraception for the duration of drug use and for 60 days after the last dose.

Exclusion Criteria:

1. Patients have a present or previous active malignancy except the diagnosis of rectal cancer this time;
2. Patients underwent major surgery within 4 weeks prior to study treatment;
3. Patients have any condition affects the absorption of capecitabine through gastrointestinal tract;
4. Patients have severe uncontrolled recurrent infections, or other severe uncontrolled concomitant diseases;
5. Patients who are allergic to any of the ingredients under study;
6. Patients with severe concomitant diseases with estimated survival ≤ 5 years;
7. Patients with present or previous moderate or severe liver and kidney damage presently or previously;
8. Patients have received other study medications or any immunotherapy currently or in the past;
9. Patients preparing for or previously received organ or bone marrow transplant;
10. Patients who received immunosuppressive or systemic hormone therapy for immunosuppressive purposes within 1 month prior to the initiation of study therapy;
11. Patients with congenital or acquired immune deficiency (such as HIV infection);
12. If patients with a history of uncontrolled epilepsy, central nervous system disease or mental disorder, the investigator will determine whether the clinical severity prevents the signing of informed consent or affects the patient's oral medication compliance;
13. Patients with other factors that may affect the study results or cause the study to be terminated midway, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring combined treatment and severe laboratory examination abnormalities.
14. Pregnant or lactating women

Criteria for Withdrawal:

1. The subject withdraws informed consent;
2. The subject requests to withdraw from the study, or loses follow-up;
3. The subject demonstrates poor compliance and is unable to participate in the treatment and visits as required by the study protocol;
4. The subject experiences intolerable adverse events, and the investigator determines that continuing the study may be detrimental to the subject;
5. Other reasons, where the investigator determines it is not suitable for the subject to continue in the study.

Criteria for Study Termination:

1. There are major errors in the study protocol;
2. The study involves significant risks and is terminated following review by the ethics committee;
3. Termination requested by the sponsor or regulatory authorities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
CR rate | from preoperative to 10 days postoperative
  complete response rate, If patients achieved cCR after neoadjuvant therapy or were confirmed pCR after TME, they were considered as complete response (CR). pCR was defined as no residual tumor cells on the histologic examination of surgical specimens according to AJCC 8th edition. cCR was defined according to the Memorial Sloan Kettering Cancer Center (MSKCC) standard.

SECONDARY OUTCOMES:
TRAE | from commencing of treatment to the 30th day after surgery
  incidence of treatment-related adverse event
30-day incidence of postoperative complications | within 30 days after surgery
  incidence of surgical complications within 30 days after surgery
ORR | before surgery
  objective response rate; The ORR rate is the result of complete response (CR) rate plus partial response (PR) rate.
3-y DFS rate | 3 years
  3-year disease free survival rate
NAR score | within 10 days after surgery
  neoadjuvant rectal score
R0 resection rate | within 10 days after surgery
  rate of R0 resection
anal preservation rate | instantly after surgery
  proportion of patients with preserved anal sphincter

OTHER OUTCOMES:
The expression of CD68 | up to 3 months after surgery
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC
The expression of CD86 | up to 3 months after surgery
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC
The expression of CD163 | up to 3 months after surgery
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC
The expression of CD4 | up to 3 months after surgery
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC
The expression of CD8 | up to 3 months after surgery
  The density, H-score of each marker in paraffin-embedded tissue sections detected by mIHC

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Friendship Hospital,Capital Medical University, Beijing
  - Peking Union Medical College Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No
Export of individual patient data is a sensitive issue according to current Chinese laws.

REFERENCES:
- [Background] Amin, M. B. et al. AJCC cancer staging manual. (New York: Springer. 252-274 2017)
- [Background] Andre T, Shiu KK, Kim TW, Jensen BV, Jensen LH, Punt C, Smith D, Garcia-Carbonero R, Benavides M, Gibbs P, de la Fouchardiere C, Rivera F, Elez E, Bendell J, Le DT, Yoshino T, Van Cutsem E, Yang P, Farooqui MZH, Marinello P, Diaz LA Jr; KEYNOTE-177 Investigators. Pembrolizumab in Microsatellite-Instability-High Advanced Colorectal Cancer. N Engl J Med. 2020 Dec 3;383(23):2207-2218. doi: 10.1056/NEJMoa2017699. PMID 33264544
- [Background] King RS, Tuthill C. Evaluation of thymosin alpha 1 in nonclinical models of the immune-suppressing indications melanoma and sepsis. Expert Opin Biol Ther. 2015;15 Suppl 1:S41-9. doi: 10.1517/14712598.2015.1008446. Epub 2015 Feb 2. PMID 25643200
- [Background] Danielli R, Cisternino F, Giannarelli D, Calabro L, Camerini R, Savelli V, Bova G, Dragonetti R, Di Giacomo AM, Altomonte M, Maio M. Long-term follow up of metastatic melanoma patients treated with Thymosin alpha-1: investigating immune checkpoints synergy. Expert Opin Biol Ther. 2018 Jul;18(sup1):77-83. doi: 10.1080/14712598.2018.1494717. PMID 30063847
- [Background] Renga G, Bellet MM, Pariano M, Gargaro M, Stincardini C, D'Onofrio F, Mosci P, Brancorsini S, Bartoli A, Goldstein AL, Garaci E, Romani L, Costantini C. Thymosin alpha1 protects from CTLA-4 intestinal immunopathology. Life Sci Alliance. 2020 Aug 14;3(10):e202000662. doi: 10.26508/lsa.202000662. Print 2020 Oct. PMID 32817121